CLINICAL TRIAL: NCT06815276
Title: Core Stability and Performance: A Randomized Control Trial in Amateur Football Players
Brief Title: Core Stability Training and Athletic Performance in Amateur Footballers
Acronym: KICK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cooperativa de Ensino Superior, Politécnico e Universitário (Other)
Responsible Party: Principal Investigator, Maria Paço, Principal investigator, Cooperativa de Ensino Superior, Politécnico e Universitário
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Core stability and performance
Record Dates: First submitted 2025-01-20; First posted 2025-02-07 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Performance; football; core; balance; agility; power
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Regular training + Core muscle training
  Interventions: Other: Exercise
- Control (No Intervention): Regular training

INTERVENTIONS:
Other: Exercise — core muscle training
  Arms: Experimental

SUMMARY:
This study aims to evaluate the effects of a core strengthening program on the athletic performance of amateur football players aged 18 to 35. Conducted as a double-blind randomized controlled trial, the research compares two groups: one undergoing traditional football training combined with a 12-week core strengthening program, and another following only regular training and matches.

Key outcomes include:

Core strength (measured using the Plank Endurance Test), Balance (assessed through the Y-Balance Test), Functional power (evaluated with the Vertical Jump Test), Overall Athletic Performance: Illinois (assessed through Illinois Agility Test)

Participants will be randomly assigned to either the experimental or control group. Assessments will be conducted pre- and post-intervention to determine the program's impact on physical fitness and performance. The findings will provide insights into whether targeted core training enhances key physical attributes and athletic abilities, critical to injury prevention, functional capacity, and athletic performance.

DETAILED DESCRIPTION:
This study will investigate the effects of a core strengthening program on the physical fitness and athletic performance of amateur football players aged 18 to 35. Designed as a double-blind randomized controlled trial, the research aims to provide robust evidence on how targeted core training influences key performance indicators, offering practical applications for physiotherapy, sports science, and athletic training.

Study Purpose

Core muscles play a pivotal role in stabilizing the spine, transferring forces, and enhancing movement efficiency during athletic activities. Weakness or instability in the core can lead to suboptimal performance and increase the risk of injuries, particularly in sports like football, where balance, agility, and power are essential. This study seeks to evaluate whether a structured, evidence-based core strengthening program can enhance core strength, balance, functional power, and overall athletic performance in amateur football players.

Methodology

A total of 50 male amateur football players from local clubs will be invited to voluntarily participate in the study. Participants will be randomly divided into two groups:

Experimental Group: Traditional football training combined with a 12-week core strengthening program.

Control Group: Followed only regular football training. The core strengthening program, inspired by McGill's principles of core training, includes progressive exercises performed three times per week for 12 weeks. Each session will last 15 minutes and will be integrated into the players' regular training schedules.

Assessments

Participants will perform comprehensive evaluations at the beginning and end of the study to measure the following outcomes:

Core Strength: Plank Endurance Test, a validated measure of muscular endurance. Balance: Evaluated with the Y-Balance Test, to assess dynamic balance and agility.

Functional Power: Measured using the Vertical Jump Test, to evaluate lower limb strength and explosive power.

Overall Athletic Performance: Illinois Agility Test, to assess agility..

Expected Impact

The findings are expected to highlight the effect of targeted core training in optimizing physical performance. This study underscores the importance of core stability as a foundational component of athletic conditioning, offering practical applications for physiotherapists, sports scientists, coaches, and athletes aiming to enhance performance and maintain physical health.

ELIGIBILITY:
Inclusion Criteria:

* Male amateur football players aged between 18 and 35 years,
* Active members of local football clubs;
* Medically cleared and physically fit to participate in regular training sessions and matches.

Exclusion Criteria:

* Individuals already engaged in a core strengthening program;
* Participants with injuries or medical conditions that contraindicate participation in the study or could interfere with the intervention.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Core Strength - Plank Endurance Test | baseline and 12 weeks
  Participants assume a prone position, supporting their body weight on forearms and toes, maintaining a straight line from head to heels. The duration for which the position is held without compromising form is recorded, reflecting the endurance capacity of the core musculature.
Balance - Y balance test | baseline and 12 weeks
  Assesses dynamic balance by having participants reach as far as possible in multiple directions with one foot while maintaining balance on the other, providing insight into lower limb stability and control.
Overall Athletic Performance - Illinois Agility Test | baseline and 12 weeks
  Measures agility by timing participants as they navigate a predetermined course involving directional changes, reflecting their ability to accelerate, decelerate, and change direction efficiently.
Functional Power: Vertical Jump Test | baseline and 12 weeks
  Participants perform a maximal vertical jump from a standing position, with the jump height measured to evaluate lower body explosive power.

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Paço, PhD, Principal Investigator — H²M - Health and Human Movement Unit, Polytechnic University of Health, CESPU, CRL 4760-409 Vila Nova de Famalicão.; Paula D Chaves, PhD, Principal Investigator — H²M - Health and Human Movement Unit, Polytechnic University of Health, CESPU, CRL 4760-409 Vila Nova de Famalicão.
Locations (1):
- Escola Superior de Saúde do Vale do Ave, Vila Nova de Famalicão, Braga District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
Deciding whether to share Individual Participant Data (IPD) involves weighing several considerations... we have to further reflect to make an informed decision about sharing IPD, balancing the potential benefits to the scientific community with the responsibility to protect participant rights and data integrity.